CLINICAL TRIAL: NCT05773261
Title: Modern Surfaces of the Uncemented Cup in Total Hip Arthroplasty: A Randomized, Clinical Investigation Comparing Two Different Ultra-porous Coated Surfaces of Uncemented Cups Using CT-based Micromotion Analysis and Clinical Evaluation
Brief Title: Clinical Investigation Comparing Two Different Ultra-porous Coated Surfaces of Uncemented Cups
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: University Hospital, Umeå (Other); Region Västerbotten (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TrabecuLINK study
Record Dates: First submitted 2022-11-21; First posted 2023-03-17 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Osteoarthritis, Hip
Keywords: Osteoarthritis; Total hip arthroplasty; Uncemented total hip arthroplasty
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Control: Pinnacle Gription series 100 cup with a Marathon liner combined med with a Corail femoral stem.
  Investigational device: MobilLINK TrabecuLINK cup with X-LINKed liner combined with a LCU femoral stem.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MobilLINK TrabecuLINK cup (Active Comparator): The investigational device in this study is the newly developed MobilLINK TrabecuLINK cup. It will in this study be combined with a uncemented LCU stem.
  The MobilLINK TrabecuLINK cups are made from Tilastan, a Ti6A4V alloy. The MobileLINK press-fit shells are hemispheric and polar flattened. An equatorial press-fit is built into the shells for primary stability after cementless implantation. All shells have a polar hole, which is used to connect an impactor handle for implantation of the shell. This polar hole can be closed with a polar screw. The MobileLINK TrabecuLINK shells have a 3D printed trabecular surface structure with a pore size of 610 to 820 μm and a porosity of 70 %.
  Interventions: Device: MobilLINK TrabecuLINK cup
- Pinnacle Gription Series 100 cup (Active Comparator): For the control group a Pinnacle Gription cup series 100 with a apex hole eliminator will be used together with a neutral cross-linked polyethylene (XLPE) Marathon liner (DePuy Synthes by Johnson & Johnson, Norderstedt, Germany). The Pinnacle Gription cup is a hemispherical, single-geometry, titanium press-fit cup with a solid body. The outer surface consists of a porous coating with 300 μm sintered titanium beads coated with an extra layer of irregularly shaped pure titanium pieces. In cases where no initial stability can be reached when using the Pinnacle 100 series, the Pinnacle Gription sector cup with additional bone screws will be used. The cross-linked Marathon insert is made of 1050 GUR resin, irradiated with 50 kGy, remelted and plasma sterilized.
  The Pinnacle Gription cup will be implanted together with a Corail stem (DePuy Synthes).
  Interventions: Device: Pinnacle Gription cup

INTERVENTIONS:
Device: MobilLINK TrabecuLINK cup — THA with MobilLINK TrabecuLINK cup and LCU stem
  Arms: MobilLINK TrabecuLINK cup
Device: Pinnacle Gription cup — THA with Pinnacle Gription cup and Coral stem
  Arms: Pinnacle Gription Series 100 cup

SUMMARY:
A randomised controlled study comparing two types of ultra-porous coated uncemented cups in total hip arthroplasty. Primary objective is to investigate if the clinical, radiological and patient-reported outcome of the new MobileLINK TabecuLINK cup combined with an X-LINKed insert is non-inferior to the clinical and radiological outcome of the Pinnacle Gription series 100 cup combined with the Marathon liner. Patients are evaluated up to 15 years postoperatively.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the clinical outcome and long-term risk of development of osteolysis of a newly introduced cementless press-fit acetabular cup, consisting of a shell with a 3D surface structure and a highly cross-linked liner by precise measurement of early migration and wear.

Migration describes the movement between the implant and the surrounding bone over time. Early migration of the implant, within 2 years after operation, has shown to be a strong predictor for increased risk for late failure. Thus, high precision migration studies can be used to evaluate the performance of new implants in small groups of patients with a relatively short observation time. Wear particles are one of the main causes of periprosthetic osteolysis. Although modern, more wear resistant materials, appears to have a greatly reduced risk of osteolysis, the desired complete elimination of osteolysis appears to be yet unachieved. It is most likely that the mechanism of periprosthetic osteolysis is multifactorial.

In this study the investigators plan to include 70 patients that are planned for operation with an uncemented total hip arthroplasty. 35 patients will be randomized to receive the new implant and 35 patients will be included in the control group and receive a standard uncemented prosthesis. All patients will then be followed with CT scans and patient reported outcome measures 3-month, 1 year, 2 years, 5 years and 15 years after the operations. The CT scans will be used both for measurement of migration and wear and development of osteolysis around the implant.

ELIGIBILITY:
Inclusion Criteria:

* Patients are foreseen for implantation of an uncemented acetabular press-fit cup and an uncemented stem
* Age 30-70 years
* Primary osteoarthritis of the hip
* Body Mass Index between 18 and 35 kg/m2
* Willingness and ability to follow clinical investigation protocol

Exclusion Criteria:

* Grossly abnormal hip anatomy (hip dysplasia, Crowe Grade 2 or above, Perthes or other causes)
* Osteoporosis
* Paget's disease
* Inflammatory arthritis
* Secondary osteoarthritis
* Presence of malignancy in the area of surgery
* Treatment with bisphosphonates, cortisol or cytostatic drugs 6 months or less prior to surgery
* Previous surgery in the affected hip
* Inclusion of the contralateral hip in this clinical investigation
* Not suited for the clinical investigation for other reason (surgeon's judgment)
* Pregnant or breastfeeding women
* Prison inmate

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-09-09 (Actual); Primary Completion 2026-09-09 (Estimated); Study Completion 2039-09-09 (Estimated)

PRIMARY OUTCOMES:
Early migration of the cup | 2 years after operation
  Migration of the cup between 3 month and 2 years after implantation of the cup measured with Computed Tomography scan based Micromotion Analysis (CTMA) in mm.

SECONDARY OUTCOMES:
Proximal wear | 5 years after operation
  Liner wear measured as proximal penetration of the femoral head prosthesis into the liner between 1 year and 5 years after operation in mm
3D wear | 5 years after operation
  Liner wear measured as 3D penetration of the femoral head prosthesis into the liner between 1 year and 5 years after operation in mm
Long term migratio | 15 years after operation
  Migration of the cup measured in mm with CTMA
Long term wear | 15 years after operation
  Liner wear measured in mm with CTMA
Stem migration | 15 years
  Distal and 3D migration in mm of the stem between post- operative examination and 3 month, 3 month and 2 years, 3 month and 5 years and 3 month and 15 years.
Patient reported outcome with Forgotten Joint Score | 15 years after operation
  Patient-reported outcome measured by Forgotten Joint Score (FSJ). The scores will be summarized and transformed to a scale ranging from 0 to 100, where a high value indicate that the patient tends to be less aware of the affected joint when performing daily activities.
Patient reported outcome with Hip dysfunction and Osteoarthritis Outcome Score | 15 years after operation
  Patient-reported outcome measured by Hip dysfunction and Osteoarthritis Outcome Score (HOOS). Each of the 5 subscales will get a score of 0 to 100, with 0 indicating extreme symptoms and 100 indicating no symptoms. The subscales will be plotted as a HOOS profile, by connecting the mean scores for all 5 dimensions with a line.
Patient reported outcome with University of California, Los Angeles Activity Score | 15 years after operation
  Patient-reported outcome measured by University of California, Los Angeles Activity Score (UCLA). The patients physical activity level rank from 1 (low) to 10 (high).
Patient reported outcome with EuroQuol 5. | 15 years after operation
  Patient reported health related quality of life, measured by EuroQuol 5 dimensions (EQ-5D). For the calculation of the EQ-5D index the standard value set version 2.1 for Sweden is used. Index scores range from 0 ( 0 is the value of a health state equivalent to dead; negative values representing values as worse than dead) to 1 (the value of full health), with higher scores indicating higher health utility.
Reoperations | 15 years after operation
  Incidence and rate of revisions, re-operations and operation-related complications
Osteolysis | 15 years after operation
  Incidence and rate of patients showing osteolysis around the cup on CT scans and/or on x-rays
Precision of migration measurements with CTMA | 1 year after operation
  Precision of migration measurement in mm with CTMA, by comparing double CT scans obtained on the same day at the 1 year follow-up.
Precision of wear mearurements with CTMA | 1 year after operation
  Precision of wear measurement in mm with CTMA, by comparing double CT scans obtained on the same day at the 1 year follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Volker Otten, M.D, PhD, Principal Investigator — Umeå University hospital/Umeå University
Locations (1):
- Volker Otten, Umeå, Västerbotten County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Buttaro MA, Onativia JI, Slullitel PA, Andreoli M, Comba F, Zanotti G, Piccaluga F. Metaphyseal debonding of the Corail collarless cementless stem: report of 18 cases and case-control study. Bone Joint J. 2017 Nov;99-B(11):1435-1441. doi: 10.1302/0301-620X.99B11.BJJ-2017-0431.R1. PMID 29092981
- [Background] Louboutin L, Viste A, Desmarchelier R, Fessy MH. Long-term survivorship of the Corail standard stem. Orthop Traumatol Surg Res. 2017 Nov;103(7):987-992. doi: 10.1016/j.otsr.2017.06.010. Epub 2017 Aug 1. PMID 28778624
- [Background] van der Voort P, Pijls BG, Nieuwenhuijse MJ, Jasper J, Fiocco M, Plevier JW, Middeldorp S, Valstar ER, Nelissen RG. Early subsidence of shape-closed hip arthroplasty stems is associated with late revision. A systematic review and meta-analysis of 24 RSA studies and 56 survival studies. Acta Orthop. 2015;86(5):575-85. doi: 10.3109/17453674.2015.1043832. PMID 25909455
- [Background] Bitsch RG, Loidolt T, Heisel C, Ball S, Schmalzried TP. Reduction of osteolysis with use of Marathon cross-linked polyethylene. A concise follow-up, at a minimum of five years, of a previous report. J Bone Joint Surg Am. 2008 Jul;90(7):1487-91. doi: 10.2106/JBJS.F.00991. PMID 18594097
- [Background] Campbell D, Mercer G, Nilsson KG, Wells V, Field JR, Callary SA. Early migration characteristics of a hydroxyapatite-coated femoral stem: an RSA study. Int Orthop. 2011 Apr;35(4):483-8. doi: 10.1007/s00264-009-0913-z. Epub 2009 Dec 13. PMID 20012862
- [Background] Goriainov V, Jones A, Briscoe A, New A, Dunlop D. Do the cup surface properties influence the initial stability? J Arthroplasty. 2014 Apr;29(4):757-62. doi: 10.1016/j.arth.2013.07.007. Epub 2013 Nov 22. PMID 24269067
- [Background] Drobniewski M, Borowski A, Synder M, Sibinski M. Results of total cementless hip joint arthroplasty with Corail stem. Ortop Traumatol Rehabil. 2013 Jan-Feb;15(1):61-8. doi: 10.5604/15093492.1032797. PMID 23510822